CLINICAL TRIAL: NCT00004137
Title: Phase II Trial of Paclitaxel, Carboplatin and Topotecan With G-CSF in Untreated Patients With Extensive Small Cell Lung Cancer
Brief Title: S9914: Combination Chemotherapy Plus Filgrastim in Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067367; S9914 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-12-10; First posted 2004-04-12 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus filgrastim in treating patients who have previously untreated extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the survival and response rate of patients with previously untreated extensive stage small cell lung cancer treated with paclitaxel, carboplatin, topotecan, and filgrastim (G-CSF). II. Determine the side effects and toxicity of this regimen in these patients.

OUTLINE: Patients receive topotecan IV over 30 minutes on days 1-4 and paclitaxel IV over 1 hour followed by carboplatin IV over 1 hour prior to topotecan on day 4. Patients receive filgrastim (G-CSF) subcutaneously once daily beginning on day 5 and continuing until blood counts recover. G-CSF must be discontinued at least 24 hours prior to beginning each subsequent course of chemotherapy. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven, previously untreated extensive stage small cell lung cancer (SCLC) Brain metastases allowed if: Asymptomatic OR Previously treated with radiotherapy and/or surgery Measurable or evaluable disease outside the area of prior surgical resection or a new lesion must be present

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than ULN Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any stage I or II cancer that is in complete remission

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior systemic biologic therapy for SCLC Chemotherapy: No prior systemic chemotherapy for SCLC Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy for SCLC Surgery: See Disease Characteristics At least 2 weeks since prior thoracic or other major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 1999-10; Primary Completion 2004-03 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dunphy, MD, Study Chair — Duke Cancer Institute
Locations (85):
- United States (85):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Hesketh PJ, McCoy J, Dunphy FR 2nd, Bearden JD 3rd, Weiss GR, Giguere JK, Atkins JN, Dakhil SR, Kelly K, Crowley JJ, Gandara DR. Phase II trial of paclitaxel, carboplatin, and topotecan with G-CSF support in previously untreated patients with extensive stage small cell lung cancer: Southwest Oncology Group 9914. J Thorac Oncol. 2006 Nov;1(9):991-5. PMID 17409984
- [Result] Dunphy F, Hesketh P, Chansky K, et al.: Southwest Oncology Group trial (SWOG) 9914: phase II trial of paclitaxel, carboplatin and topotecan (PCT) in untreated patients (pts) with extensive small cell lung cancer (SCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1184, 2002.